CLINICAL TRIAL: NCT06883045
Title: A Novel mHealth Intervention to Improve Outcomes of Children With Medical Complexity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Flory Nkoy, Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00179595; 1R01NR020784-01A1 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Children With Medical Complexity

STUDY DESIGN:
Intervention Model Description: We will assess the efficacy MyChildCMC app in a 6-month, 2-arm (MyChildCMC vs usual care) trial of Children with Medical Complexity (CMC) of ages between 1-18 years and their parents. Parents assigned to MyChildCMC will use the app daily for 6 months to monitor their vital signs/symptoms. Those assigned to usual care will use a paper diary for 6 months to monitor their vital signs/symptoms. Both arms will receive financial incentive for daily monitoring (monitoring incentive) and for responding to surveys.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyChildCMC group (Experimental): MyChildCMC is an app designed to support remote monitoring of CMC crosscutting symptoms to identify signs of CMC's health deterioration early to change their care early to avoid progression and prevent ED/hospital admissions. The app includes the following features: 1) automated reminders, 2) vital sign/symptom monitoring, 3) real-time feedback system, 4) automated and real-time summary reports with longitudinal graphs, 5) automated alerts to a care coordinator, and 6) clinic dashboard connecting patients to clinics and allowing access to patient data to support care coordination. Those randomized to MyChildCMC will use the app daily for 6 months to monitor vital signs/symptoms. They will also receive a sensor (Masimo Mighty Sat) to facilitate collection of Oxygen saturation, heart rate and respiratory rate, as well as financial incentive for daily monitoring (monitoring incentive) for 6-months and for responding to surveys.
  Interventions: Other: MyChildCMC app (an app designed to facilitate home monitoring of CMC's health status)
- Usual care group (Active Comparator): Those assigned to usual care will use a paper diary to monitor their vital signs and symptoms daily for 6 months. They will also receive a sensor (Masimo Mighty Sat) to facilitate collection of Oxygen saturation, heart rate and respiratory rate, as well as financial incentive for daily monitoring (monitoring incentive) for 6-months and for responding to surveys.
  Interventions: Other: MyChildCMC app (an app designed to facilitate home monitoring of CMC's health status)

INTERVENTIONS:
Other: MyChildCMC app (an app designed to facilitate home monitoring of CMC's health status) — MyChildCMC is an app designed to support remote monitoring of CMC crosscutting symptoms to identify signs of CMC's health deterioration early to change their care early to avoid progression and prevent ED/hospital admissions. The app includes the following features: 1) automated reminders, 2) vital sign/symptom monitoring, 3) real-time feedback system, 4) automated and real-time summary reports with longitudinal graphs, 5) automated alerts to a care coordinator, and 6) clinic dashboard connecting patients to clinics and allowing access to patient data to support care coordination.

SUMMARY:
Children with medical complexity (CMC) are the most vulnerable of children with chronic diseases, who have complex, multisystem chronic diseases affecting ≥3 organ systems, severe functional limitations and technology dependencies. CMC have high health care needs, and account for 40% of hospitalized children and 35% of all pediatric health care costs. Due to high medical fragility, CMC have frequent acute deteriorations superimposed on their chronic conditions, leading to recurrent emergency department (ED)/hospital admissions and affecting quality of life (QOL). To reduce ED/hospital admissions for CMC, remote monitoring is suggested, with use of mHealth apps to regularly assess their health status remotely and identify early signs of acute deterioration, allowing for early interventions to prevent ED/hospital admissions. Yet no app to support remote monitoring of CMC exists. Variable, multisystem conditions among CMC make it difficult to develop an app. Also, many CMC are at high-risk for health care inequities, with minorities having higher unmet needs, but the impacts of health care inequities and social determinants of health (SDOH) on ED/hospital admissions in CMC are rarely studied. Fortunately, ED/hospital admissions for CMC are often preceded by a limited set of shared (crosscutting) acute symptoms. These crosscutting symptoms rarely occur suddenly. Studies suggest that they usually start as subtle signs, often unnoticed by parents until they escalate to prompt an ED/hospital visit. Thus, crosscutting symptoms offer an opportunity for a novel and practical approach for developing a remote monitoring app for CMC, despite their multiple, variable underlying conditions. In a focus group, parents identified the crosscutting symptoms that most often preceded their children's hospital admissions, and conveyed their needs, preferences and key functionalities that led to MyChildCMC, the first app designed to monitor and identify early signs of crosscutting symptoms in CMC. In a pilot trial of 50 subjects, we confirmed feasibility of MyChildCMC use by parents, ability to detect early signs 2-14 days prior to ED/hospital admissions, and use leading significantly to fewer hospital days than controls. The current study will assess the efficacy and sustainability of MyChildCMC in a fully-powered 6-month, 2-arm (MyChildCMC vs usual care) trial of CMC (age 1-18 years) and their parents. Parents assigned to MyChildCMC will use the app daily for 6 months, both arms will receive financial incentive for participation, then we will stop the incentive and follow subjects for 6 more months to assess sustainability at 12 months. We will also assess if MyChildCMC use will help reduce or eliminate inequities in ED/hospital admissions. Specific Aims are: 1) Determine MyChildCMC's efficacy on 1.a. Child (ED/hospital use, hospital days and QOL) and 1.b. Parent (satisfaction, self-efficacy and stress) outcomes; 2) Compare ED/hospital use among racial/ethnic and SDOH subgroups to assess potential effect of MyChildCMC on inequities.

DETAILED DESCRIPTION:
Children with medical complexity (CMC) have complex, multisystem chronic diseases, neurological impairments with marked intellectual/physical disabilities, functional limitations, technology dependencies, high medical fragility, and account for 35% of all pediatric US health care costs. Compared to typically developing children, CMC have frequent acute health deteriorations, leading to recurrent emergency department (ED)/hospital visits.

CMC have significant daily care needs, requiring continuous care at home and substantial care coordination. Care coordination programs exist to support CMC's daily care needs, including medical homes, home health care, hospital-to-home transition, and complex care services. Observational studies of these programs report some reductions in admissions, length of stay and costs. Despite these care coordination programs, CMC continue to have frequent acute deteriorations of their health that affect their quality of life (QOL) and lead to recurrent ED/hospital admissions, many of which are avoidable with early detection and intervention.

Remote monitoring with support of mHealth apps has been suggested to improve CMC care, QOL, and help reduce their ED/hospital admissions. This can be done via regular assessment of CMC's health status and detection of early signs of deteriorations to prompt early interventions. Unfortunately, no remote monitoring app for CMC exists. Available remote monitoring apps target primarily non-complex single chronic conditions (e.g. asthma, diabetes). Variable, multisystem conditions make it difficult to develop a remote monitoring app for CMC.

ED/hospital admissions for CMC are often preceded by a limited set of shared (crosscutting) acute symptoms: fever, respiratory distress with decreased oxygenation, feeding/fluid intolerance, altered mental status (sometimes seizures), and pain. These symptoms rarely occur suddenly. Studies suggest that they usually start as subtle signs (e.g. change in vital signs), often unnoticed by parents until they escalate to prompt an ED/ hospital visit. Thus, crosscutting symptoms provide an opportunity for a novel and practical approach for remote monitoring. In a focus group we conducted, CMC parents identified these crosscutting symptoms preceding most of their CMC's admissions. They also conveyed their needs, preferences and key functionalities that led to MyChildCMC, the first app for CMC remote monitoring, which has: 1) automated daily reminders, 2) crosscutting symptom monitoring, 3) automated feedback, 4) automated reporting with graphs, and 5) automated alerts.

In a 3-month pilot trial of 50 CMC randomized to MyChildCMC (n=24) or usual care (n=26) our team conducted, MyChildCMC use by parents showed high feasibility (high participation, adherence and retention), ability to detect early signs of crosscutting symptoms 2-14 days prior to most ED/hospital admissions, fewer hospital days, and higher parent satisfaction than controls. But, MyChildCMC's efficacy for ED/hospital admissions has yet to be demonstrated in a fully powered study (pilot was not powered for number of ED/hospital admissions).

The proposed multicenter study will test MyChildCMC's efficacy in a 6-month trial in which 360 CMC (age 1-18 years) and parents will be randomly assigned to MyChildCMC or usual care. Both groups will receive financial incentive for participating. Those randomized to MyChildCMC will use the app daily for 6 months to monitor their child's crosscutting symptoms and receive immediate feedback. Alerts for early signs of deteriorating CMC's health will be sent to parents, and their clinic care coordinators (or heath care providers) for follow-up. At end of 6 months, we will stop the incentive and follow subjects for 6 more months to assess sustainability at 12 months.

We will also assess if MyChildCMC use helps reduce or eliminate inequities in ED/hospital admissions. CMC are at-risk for inequities as many CMC families report higher financial and social hardships, with minorities having higher unmet needs. Continuous attention to CMC's medical needs and caregiving can lead to high parental stress. Recurrent health deteriorations and admissions contribute to parent work disruptions, work loss, and poverty, compromising family's wellbeing. Though social determinants of health (SDOH) contribute to health inequities, impacts of apps on SDOH inequities in CMC have not been studied. Our Specific Aims are:

Aim 1: Determine MyChildCMC's impact on 1.a. Child (ED/hospital use, hospital days and QOL) and 1.b. Parent (satisfaction, self-efficacy and stress) outcomes. H1. MyChildCMC users will have less ED/hospital use and hospital days, higher child's QOL, higher satisfaction, higher caregiving self-efficacy, and lower stress.

Aim 2: Compare ED/Hospital use among racial/ethnic and SDOH subgroups to assess potential effect of MyChildCMC on inequities. H2: ED/Hospital use will be reduced with MyChildCMC use vs controls in each subgroup, and inequities eliminated in racial/ethnic minority/disadvantaged subgroups with high use adherence.

Significance: Our study is based on promising pilot data supporting the feasibility of CMC remote monitoring. If efficacious, it will be a new model for improving care, reducing/eliminating inequities in disadvantaged subgroups and reducing ED/Hospital admissions in CMC, generalizable to all children with multiple chronic conditions.

ELIGIBILITY:
Inclusion Criteria:

* CMC, ages 1-18 years and their parents (or primary caregivers)
* CMC (inpatients or outpatients) who receive care at participating sites (comprehensive care clinics for CMC)
* Own (or provided) a smartphone or tablet with internet access
* Speak English or Spanish.
* CMCs are identified using an operational definition, as having: 1) multisystem chronic diseases involving ≥3 organ systems, 2) ≥3 HCPs involved in their care, 3) high fragility or frequent (≥2) or 1 prolonged (>10 days) hospitalization in the prior year, and/or 4) medical technology dependence.

Exclusion Criteria:

* Critically ill CMC and infants.
* CMC exhibit similar developmental and functional abilities and typically function below expected for a 7-year-old child, allowing inclusion of a wide age range in studies.
* Infants were excluded as many CMC <1 year have prematurity-related conditions that may resolve by age 2.
* CMC >18 years of age were not included as some may transition to adult health care.
* Note: No one will be excluded due to lack of smartphone/internet access. We estimated <10% of families may not have a smartphone/internet, and will provide them low-cost tablets and cellular internet access.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 360 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
ED/hospital admissions | 6-month pre and 6-month post enrollment
  Numbers of ED and hospital admissions will be assessed pre-post enrollment.

SECONDARY OUTCOMES:
Child's quality of life (QOL) | Baseline, 1 month, 3 months and 6 months post-enrollment
  Child's QOL will be assessed using a survey CMC specific survey questionnaire (adapted from Ellzey et al.). This is a 7-item survey questionnaire that assesses physical health, mental health, sleep, pain, activities, and general QoL. The total QoL score will be standardized to 100 points, with highest (100) reflecting the best QOL.
Self-efficacy scale | Baseline, 1 month, 3 months and 6 months post-enrollment
  Caregiving self-efficacy will be collected using a CMC specific questionnaire adapted from validated surveys, including the PROMIS and PhenX Toolkit self-efficacy scales, as no existing scale meets CMC needs. This is a 10-item questionnaire with scores ranging from 10 (lowest self-efficacy) to 50 (highest self-efficacy).
Caregiver stress | Baseline, 1 month, 3 months and 6 months post-enrollment
  Caregiver stress will be assessed using the Short Form Zarit Burden Interview (ZBI-12). The ZBI-12 is a self-administered 12-item validated survey, with 5 responses ranging from 0 (never) to 4 (always), and a total score rating care-giving stress from 0 (no stress) to 48 (high/severe stress).
Parent satisfaction | Baseline and 6 months post-enrollment
  Parent satisfaction will be collected using the Client Satisfaction Questionnaire. This is a 7-item questionnaire that assesses parent satisfaction with the child health care, with total scores ranging from 7 (lowest satisfaction) to 35 (highest satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Flory Nkoy, MD, MS, MPH, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nkoy F, Stone B, Hofmann M, Fassl B, Zhu A, Mahtta N, Murphy N. Home-Monitoring Application for Children With Medical Complexity: A Feasibility Trial. Hosp Pediatr. 2021 May;11(5):492-502. doi: 10.1542/hpeds.2020-002097. Epub 2021 Apr 7. PMID 33827786
- [Background] Nkoy FL, Hofmann MG, Stone BL, Poll J, Clark L, Fassl BA, Murphy NA. Information needs for designing a home monitoring system for children with medical complexity. Int J Med Inform. 2019 Feb;122:7-12. doi: 10.1016/j.ijmedinf.2018.11.011. Epub 2018 Nov 26. PMID 30623786